CLINICAL TRIAL: NCT07067502
Title: Impact of Biphasic Cuirass Ventilation Compared to Non-Invasive Ventilation in High Risk Extubations
Brief Title: Impact of Biphasic Cuirass Ventilation Compared to Non Invasive Ventilation in High Risk Extubations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Hayek Medical (Unknown)
Responsible Party: Principal Investigator, Dennis Chairman, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 455329
Record Dates: First submitted 2025-06-27; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Failure; Extubation Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non Invasive ventilator arm (per current standard of care) (Active Comparator): per current standard of care
  Interventions: Device: Biphasic cuirass ventilator which is a type of negative pressure ventilator will be applied to patients on the intervention arm
- Biphasic cuirass ventilator arm (Experimental): patients in this arm will be the intervention arm and will be placed on the Biphasic cuirass ventilator.
  Interventions: Device: Biphasic cuirass ventilator which is a type of negative pressure ventilator will be applied to patients on the intervention arm

INTERVENTIONS:
Device: Biphasic cuirass ventilator which is a type of negative pressure ventilator will be applied to patients on the intervention arm — As opposed to patients being placed on Non invasive ventilation (CPAP or BiPAP) the intervention arm patients will be placed on the Biphasic cuirass ventilator which is a form of negative pressure ventilator.

SUMMARY:
subjects on mechanical ventilator who are about to be extubated to Non invasive ventilation because the physician thinks they are high risk for failure will be approached and consented for our study. Once randomized they will either be on the standard of care Non invasive arm or the intervention arm which would mean they are placed on the Biphasic cuirass ventilation.

DETAILED DESCRIPTION:
We are planning on conducting a pilot study to assess if Biphasic cuirass ventilator is non inferior to Non invasive ventilation in high risk patients who are usually extubated to Non Invasive ventilation per current standard of care.

We will identify daily in our Medical Intensive care unit patients who have passed their spontaneous breathing trials and are being planned on being extubated to Non invasive ventilation per their treating Physician and will screen them for suitability and if so then one of our study team will approach patient and or their durable power of attorney and explain about our study and possible risks vs benefit and if they are agreeable will get a written consent and then they are randomized to either the Non invasive arm (per current standard of care) vs Biphasic cuirass ventilation arm (intervention arm).

We plan on assessing them per current standard of care with blood gas and other routine standard laboratory and or imaging. The subjects will not be compensated and they will be made aware of this upfront. Also their participation is completely voluntary and they will not get any additonal charge for taking part in the study. Assuming they tolerate the biphasic cuirass ventilator we anticipate them being on it anywere from 1-4 days.

ELIGIBILITY:
Inclusion Criteria:

* High risk extubation patients in the Medical Intensive care units who are being thought to be placed on non invasive ventilator post extubation.

Exclusion Criteria:

* Age <18 or >80
* Pregnant
* Inmate/Prisoner
* Chest wall defects
* BMI >50
* History of Diaphragmatic paralysis
* History of Neuromuscular disease
* Contraindication to study device (open chest wound, flail chest, complex thoracic surgeries in the past)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
to assess for non-inferiority of Biphasic cuirass ventilator compared to Non invasive ventilator in high risk extubations. | 1 year
  Primary outcome will try to assess for non-inferiority of Biphasic cuirass ventilator compared to Non invasive ventilator in high risk extubations - In other words we are comparing and calculating the rate of re-intubations in these patients in the two arms viz. Standard of care Non Invasive Positive Pressure ventilation vs intervention arm using the Biphasic Cuirass Ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis B Chairman, MD, Principal Investigator — T

IPD SHARING:
Plan to Share IPD: No
we don't need individual personalized data as most data will be grouped in either arms and would include age sex BMI and disease condition and their personalized data are not necessary for the research paper.

REFERENCES:
- [Background] Burns KE, Meade MO, Premji A, Adhikari NK. Noninvasive positive-pressure ventilation as a weaning strategy for intubated adults with respiratory failure. Cochrane Database Syst Rev. 2013 Dec 9;2013(12):CD004127. doi: 10.1002/14651858.CD004127.pub3. PMID 24323843
- [Background] El-Solh AA, Aquilina A, Pineda L, Dhanvantri V, Grant B, Bouquin P. Noninvasive ventilation for prevention of post-extubation respiratory failure in obese patients. Eur Respir J. 2006 Sep;28(3):588-95. doi: 10.1183/09031936.06.00150705. Epub 2006 May 31. PMID 16737982
- [Background] Ferrer M, Valencia M, Nicolas JM, Bernadich O, Badia JR, Torres A. Early noninvasive ventilation averts extubation failure in patients at risk: a randomized trial. Am J Respir Crit Care Med. 2006 Jan 15;173(2):164-70. doi: 10.1164/rccm.200505-718OC. Epub 2005 Oct 13. PMID 16224108
- [Background] Nava S, Gregoretti C, Fanfulla F, Squadrone E, Grassi M, Carlucci A, Beltrame F, Navalesi P. Noninvasive ventilation to prevent respiratory failure after extubation in high-risk patients. Crit Care Med. 2005 Nov;33(11):2465-70. doi: 10.1097/01.ccm.0000186416.44752.72. PMID 16276167
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265